CLINICAL TRIAL: NCT06695286
Title: Impact of Intensive Outpatient Rehabilitation on Non-Motor Patient-Reported Outcomes in Parkinson's Disease: The INTENSO Study
Brief Title: Impact of Intensive Outpatient Rehabilitation on Non-Motor Patient-Reported Outcomes in Parkinson's Disease (INTENSO)
Acronym: INTENSO
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Marianna Capecci, PhD, Professor, Università Politecnica delle Marche
Other Study IDs: ID 101/2024, number 3054
Record Dates: First submitted 2024-11-09; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; rehabilitation; non-motor symptoms; multimodal; exercise; intensity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with Parkinson's Disease consecutively referred to the outpatient rehabilitation facility: Single center historical cohort study of people with PD consecutively referred to the outpatient rehabilitation facility of a Center for Diagnosis and Treatment of Movement Disorders, based in a university hospital in Italy.
  Interventions: Other: Multimodal rehabilitation training at high intensity; Other: Multimodal rehabilitation training at low intensity

INTERVENTIONS:
Other: Multimodal rehabilitation training at high intensity — In High Intensive Training patients received 1800 minutes of training globally.
  In our practice, a single outpatient session varies from 60 to 90 minutes, the number of sessions per cycle from 10 to 20, and the frequency from 2 days a week to 5 days a week.
  Irrespective of total course intensity, each session comprises at least 15 minutes of aerobic training (over ground or treadmill) and 10 minutes of flexibility and strengthening exercise.
  No less than 10 minutes of balance training, 10 minutes of overground training in dual tasks, and 15 minutes of occupational therapy are additionally delivered. The duration of the single training components in each session may increase according to the patients' functioning profiles, requesting a more intensive practice of gait, balance or trunk alignment or a focused training of arm dexterity or basic ADL.
Other: Multimodal rehabilitation training at low intensity — In Low Intensive Training patients received less than 900 minutes of training globally.
  In our practice, a single outpatient session varies from 60 to 90 minutes, the number of sessions per cycle from 10 to 20, and the frequency from 2 days a week to 5 days a week. Irrespective of total course intensity, each session comprises at least 15 minutes of aerobic training (over ground or treadmill) and 10 minutes of flexibility and strengthening exercise. No less than 10 minutes of balance training, 10 minutes of overground training in dual tasks, and 15 minutes of occupational therapy are additionally delivered. The duration of the single training components in each session may increase according to the patients' functioning profiles, requesting a more intensive practice of gait, balance or trunk alignment or a focused training of arm dexterity or basic ADL.

SUMMARY:
This historical cohort study aims to evaluate the impact of different intensity rehabilitation protocols on the short and medium-term severity of non-motor symptoms in patients with Parkinson's Disease. One of the principal strengths of this study is that it is a real-life study, so it has a high external validity necessary to test the clinical effectiveness of these two types of training, which could have significant practical implications for rehabilitation in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* adults diagnosed with Idiopathic PD, Hoehn & Yahr stage ≥ 1 < 5, consecutive referral to the rehabilitation facility between 1 January 2014 and 31 December 2019 to receive outpatient physiotherapy treatment for the management of motor disability, specifically targeting gait, balance, or posture disorders;
* completion of the course of rehabilitation treatment;
* availability of Non-Motor Symptom Scale and Unified Parkinson's Disease Rating Scale, recorded before and after treatment and 6 plus or minus 1 months later

Exclusion Criteria:

* diagnosis of any primary or secondary parkinsonism rather than PD
* symptom onset since less than three years
* any concomitant neurological disease (e.g. polyneuropathy, stroke, etc)
* any other chronically disabling disease (e.g. severe heart, liver or kidney failure, cancer, psychiatric disorders, limb amputation, severe musculoskeletal or neuropathic pain)
* changes in antiparkinsonian drug therapy during the whole study period
* exposure to a course of physiotherapy during the 6 months preceding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is characterized by people with Parkinson's Disease consecutively referred to the outpatient rehabilitation facility of a Center for Diagnosis and Treatment of Movement Disorders, based in a university hospital in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in Non-motor Symptoms | before treatment, immediately after treatment, and six months following the end of the treatment
  The changes in non-motor symptoms mesaured by the Non Motor Symptoms Scale ( NMSS; score range: 0-360; higher scores mean a worse outcome)
Changes in Non-motor Symptoms | before treatment, immediately after treatment, and six months following the end of the treatment
  The changes in non-motor symptoms mesaured by the Unified Parkinson's Disease Rating Scale part I ( UPDRS part I; score range 0-52; higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Changes in Parkinson's Disease related disability | before treatment, immediately after treatment, and six months following the end of the treatment
  The Parkinson's Disease related disability measured by the the Unified Parkinson's Disease Rating Scale part II (UPDRS Part II; score range 0-52; higher scores mean a worse outcome)
Changes in motor symptoms severity | before treatment, immediately after treatment, and six months following the end of the treatment
  Changes in motor symptoms severity measured by the Unified Parkinson's Disease Rating Scale part III (UPDRS Part III; score range 0-128; higher scores mean a worse outcome)
Changes in the severity of the Freezing of Gait | before treatment, immediately after treatment, and six months following the end of the treatment
  The changes in Severity of the Freezing of Gait mesaured by the Freezing of Gait Questionnaire (FOGQ; score range 0-24; higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Capecci, MD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- Department of Experimental and Clinical Medicine, Politecnica delle Marche University,, Ancona, AN, Italy